CLINICAL TRIAL: NCT04138732
Title: Health Behaviors of Medical Personnel in Hospital Maternity Ward- Community Based Participatory Pilot
Brief Title: Health Behaviors of Medical Personnel in Hospital Maternity Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 723HBM- HMO-CTIL
Record Dates: First submitted 2017-08-27; First posted 2019-10-24 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Health Behavior; Behavior
Keywords: Community; Health; Hospital
MeSH Terms: conditions — Health Behavior; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention treatment group (Experimental): This arm will receive the intervention treatment aimed to help improve their health behaviors. Interventions will include nutrition workshops and personal consultation for employees at risk, environmental intervention that includes brief exercise session prior to weekly meetings, placement of sports equipment in the department, and pedometer program, and stress reduction workshops. Healthy options will be demarcated in the hospital cafeteria.
  Interventions: Behavioral: Improve health behaviors of medical personel
- Control group (Other): This arm will be the control group and not receive the intervention treatment aimed to help improve their health behaviors.Once completing their time as the control group, they will continue into another phase of the trial and receive the intervention treatment.
  Interventions: Behavioral: Improve health behaviors of medical personel

INTERVENTIONS:
Behavioral: Improve health behaviors of medical personel — This arm will receive the intervention treatment aimed to help improve their health behaviors, as determined by employee-based steering committee. Interventions will target nutrition, physical activity and stress reduction

SUMMARY:
The purpose of this study is to characterize the existing health behaviors and obstacles to healthy lifestyle among the medical staff in a maternity ward in order to develop a specifically-tailored intervention to help improve the health behaviors of hospital shift workers.The findings will be used to establish a community-based participatory health-promoting program in the ward, engaging the staff in its development and implementation.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the existing health behaviors and obstacles to healthy lifestyle among the medical staff in a maternity ward in order to develop a specifically-tailored intervention to help improve the health behaviors of hospital shift workers. Shift-work has been associated with unhealthy lifestyles and increased risk of digestive disorders, heart conditions, various kinds of cancer, reproductive dysfunction, and mental conditions. Thus, the findings will be used to establish a community-based participatory health-promoting program in the ward, engaging the staff in its development and implementation. Community Based Participatory (CBP) approach will be used to build an evaluation and intervention. Baseline/needs assessment will be performed by mixed methods approach, combining in depth interviews with key personnel, focus groups and questionnaires that ask about demographics, physical activity and nutrition behaviors, stress, burnout, BMI, and cardiac risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Doctors, nurses, secretaries, and assistants

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiac risk factors | at the end of the 1 year treatment
  Initially assessed by in depth interviews with key personnel and focus groups and then assessed by self report through questionnaires.

SECONDARY OUTCOMES:
BMI | at the end of 1 year of treatment
  pre and post assesment of BMI via self reporting
Burnout | at the end of the 1 year treatment,
  Initially assessed by in depth interviews with key personnel and focus groups and then assessed by self report through questionnaires.
Nutrition behaviors | at the end of the 1 year treatment
  Initially assessed by in depth interviews with key personnel and focus groups and then assessed by self report through questionnaires assessing mediterrean diet adherence and western diet behavior
Physical activity minutes per week | at the end of the 1 year treatment
  Initially assessed by in depth interviews with key personnel and focus groups and then assessed by self report through questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No